CLINICAL TRIAL: NCT02885766
Title: A Multicenter, Open Label Cohort Phase 1 Dose Finding Study to Evaluate Tolerability, Safety, Pharmacokinetics and Preliminary Efficacy of PF-114 Mesylate for Oral Administration in Adult Patients With Philadelphia Chromosome Positive (Ph+) Chronic Myeloid Leukemia (CML), Which is Resistant to the 2-nd Generation Bcr-Abl Inhibitors or Has T315I Mutation in the BCR-ABL Gene
Brief Title: Study to Evaluate Tolerability, Safety, Pharmacokinetics and Preliminary Efficacy of PF-114 for Oral Administration in Adults With Ph+ Chronic Myeloid Leukemia, Which is Resistant to the 2-nd Generation Bcr-Abl Inhibitors or Has T315I Mutation in the BCR-ABL Gene
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fusion Pharma LLC (Industry)
Collaborators: OCT LLC (Industry); Data Matrix Solutions (Other); Skolkovo Innovation Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PF-114-01
Record Dates: First submitted 2016-08-03; First posted 2016-08-31 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Chronic Myeloid Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive
Keywords: CML; Myeloid leukaemia chronic; CML progression; Chronic phase chronic myeloid leukemia; PF-114; Cytogenetic response CCyR; Major molecular response MMR; Complete molecular response CMR; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; 2-nd generation Bcr-Abl inhibitors resistant
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — PF-114

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PF-114 (Experimental): PF-114 From 50 mg up to the MTD. Dose escalation for each next cohort is conducted by increasing the dose by 20 % (or the closest lower level, which is a multiple of 25 mg) if there are Grade 3 ADRs according to NCI CTC AE v.4 without reaching а MTD. An increase of the dose by 40 % is applied if there were Grade 2 ADRs. In the absence of Grade 2 or 3 ADRs an increase of 100 % is applied.
  When the dose reaches 400 mg/day, the following increase in dose can be made after discussing results of safety findings of PF-114 between the Investigators and the Sponsor.
  Orally, once daily
  Interventions: Drug: PF-114

INTERVENTIONS:
Drug: PF-114

SUMMARY:
A multicenter, open label cohort Phase 1 dose finding study to evaluate tolerability, safety, pharmacokinetics and preliminary efficacy of PF-114 for oral administration in adult patients with Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML), which is resistant to the 2-nd generation Bcr-Abl inhibitors or has T315I mutation in the BCR-ABL gene.

DETAILED DESCRIPTION:
PF-114 is a low molecular inhibitor of a Bcr-Abl kinase activity, which is active with respect to native and mutated forms of this enzyme with mutations in Abl kinase domain. Preclinical in vitro and in vivo studies have demonstrated the ability of PF-114 to inhibit wild Bcr-Abl type and with T315I mutation, as well as other kinds of Bcr-Abl with mutations in kinase domain, including combined mutations.

In contrast to ponatinib, PF-114 is being developed to increase the action selectivity with respect to Bcr-Abl, which potentially should increase safety of drug application in people. The results of performed preclinical studies confirmed improved selectivity of PF-114 action with respect to Bcr-Abl kinases as compared to ponatinib.

Indication:

Adult patients with Ph+ CML in chronic phase (CP) or accelerated phase (AP) resistant to previous treatment with at least one 2-nd generation inhibitor of Bcr-Abl (dasatinib, nilotinib, bosutinib) or intolerant of approved Bcr-Abl inhibitors or with T315I mutation in the BCR-ABL gene

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria in order to be eligible for participation in the study:

1. Able to give written informed consent;
2. Male or female patient ≥ 18 years old;
3. Confirmed diagnosis of CML in chronic or accelerated phase according to European LeukemiaNet guideline as of 2013;
4. Available information regarding resistance to the therapy with least one 2-nd generation Bcr-Abl inhibitor (dasatinib or nilotinib or bosutinib), or intolerance of approved Bcr-Abl inhibitors, or presence of T315I mutation irrespective of treatment history;
5. In case of previous history of blast crisis phase of CML at least 6 months are required to pass after the end of blast crisis phase before the first dose of PF-114;
6. ECOG performance status ≤ 2 (see Appendix 2);
7. Adequate renal function defined as serum creatinine ≤ 1.5 times upper limit of normal (ULN);
8. Adequate hepatic function defied as:

   * serum bilirubin ≤ 1.5 X ULN unless a patient is diagnosed with Gilbert's syndrome;
   * serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 X ULN;
   * alkaline phosphatase ≤ 2.5 X ULN;
   * INR ≤ 1.5 X ULN;
9. Adequate cardiac function defined as LVEF > 40 % by echocardiogram;
10. QTcF < 470 ms;
11. Patient has recovered (to Grade 1 or less according to NCI CTCAE V 4.0) from toxicities (excluding alopecia) associated with any prior treatments;
12. Female patients of childbearing potential and male patients who have female partners of childbearing potential must agree with abstinence from sexual relations or use effective methods of contraception throughout participation in the study;
13. Ability to comply with study procedures in the Investigator's opinion.

Exclusion Criteria:

Patients must not meet any of the following criteria in order to be eligible for participation in the study:

1. Use of the following previous therapy:

   1. chemotherapy ≤ 21 days (except hydroxyurea for which washout is not required) prior to the first dose of PF-114 mesylate; оr nitrosoureas оr mitomycin С ≤ 42 days prior to the first dose of PF-114 mesylate;
   2. approved tyrosine kinase inhibitors or investigational agents ≤ 4 days prior to the first dose of PF-114;
   3. radiotherapy ≤ 28 days prior to the first dose of PF-114 ;
   4. autologous оr allogeneic stem сеll transplant < 90 days prior to enrollment;
2. Significant uncontrolled cardiac disease;
3. Sustained uncontrolled hypertension ≥ Grade 2 (according to NCI CTC AE v4);
4. Patient is taking medicinal products known to prolong the QT interval on the electrocardiogram, unless they are absolutely necessary in the opinion of the investigator;
5. Evidence of on-going graft versus host disease (GVHD), or GVHD requiring immunosuppressive therapy. Patients should be off immunosuppressive therapy for prophylaxis and/or treatment for at least 14 days prior to the first dose of PF-114;
6. Major surgery within 35 days prior to enrollment;
7. Uncontrolled intercurrent illness including, but not limited to the following: active systemic infection, uncontrolled seizure disorder, psychiatric or social circumstances that would limit compliance with study requirements or misrepresent results of the study;
8. Patient is unable to swallow study drug or has gastro-intestinal disorders that could negatively affect oral absorption of PF-114 ;
9. Any malignancy other than CML within the past 3 years (except for non-melanoma skin cancer or cervical cancer in situ).
10. Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
DLTs during the first cycle of therapy | 1-st Cycle of Therapy - 28 days
  To study the dose-limiting toxicities (DLTs) of PF-114 mesylate in the target patient population during the 1-st cycle of treatment
MTD | 1-st Cycle of Therapy - 28 days
  Primary Objectives:
  To determine the maximum tolerated dose (MTD) of PF-114 in the target patient population.

SECONDARY OUTCOMES:
The incidence of AEs | through study completion, an average of 1 year
  To assess the safety and tolerability of PF-114 in the target patient population
Cmax for oral PF-114 in the target patient population | 31 days
Tmax for oral PF-114 in the target patient population | 31 days
AUC0-t for oral PF-114 in the target patient population | 31 days
AUC0-∞ for oral PF-114 in the target patient population | 31 days
T1/2 for oral PF-114 in the target patient population | 31 days
CL/F for oral PF-114 in the target patient population | 31 days
Vd/F for single and multiple dosing for oral PF-114 in the target patient population | 31 days
Ctrough for multiple dosing for oral PF-114 in the target patient population | 31 days
Hematological response to the treatment based on European LeukemiaNet criteria, 2013. | through study completion, an average of 1 year
  Hematological response is evaluated on Day 1 of each therapy cycle
  Full hematologic response:
  Leukocytes < 10 х 109 /L Basophils < 5 % Thrombocytes < 450 х 109 /L No myelocytes, promyelocyts, myeloblasts in the differential Absence of splenomegaly - spleen non palpable
Molecular response - the level of BCR-ABL transcripts in the peripheral blood, determined by the method of quantitative polymerase chain reaction (qPCR) using the international scale. | through study completion, an average of 1 year
  Molecular response is evaluated on Day 1 of Cycles 2, 4, 7, 10. For cycles > 12, the molecular response will be evaluated once in 3 months, where the procedure is carried out for the first time during Cycle 13.
Cytogenetic response evaluated using the chromosome banding method (in situ (FISH) fluorescence hybridization is allowed only if the chromosome banding method cannot provide enough information). | through study completion, an average of 1 year
  Cytogenetic response is evaluated on Day 1, Cycles 4, 7, 13. Then if the level of BCR-ABL transcripts exceeds the level of 0.1% using the qPCR method using the international scale, cytogenetic response is evaluated no earlier than in 3 months after the previous cytogenetic analysis. After the complete cytogenetic response has been reached (CCyR), cytogenetic analysis will be carried out every 12 months.

OTHER OUTCOMES:
Pharmacodynamic response criterion to PF-114 (change in the level of pCrkL in PBL during therapy compared to baseline level) | 20 months
  To assess pharmacodynamic response to PF-114 mesylate in patients who are not in complete hematologic response upon enrollment into the study by measuring the difference of pCrkL levels in peripheral blood leukocytes (PBL) during therapy compared to baseline
The number of patients who satisfy the pharmacodynamic response criterion depending on the mutation status of BCR-ABL | 20 months
The number of patients who satisfy the hematologic response depending on the mutation status of BCR-ABL | 20 months
The number of patients who satisfy the cytogenetic response depending on the mutation status of BCR-ABL | 20 months
The number of patients who satisfy the molecular response depending on the mutation status of BCR-ABL | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Turkina, Professor, Principal Investigator — Federal Haematological Scientific Center
Locations (3):
- Russia (3):
  - Federal Haematological Scientific Center, Moscow
  - Moscow City Centre of Hematology based on City Hospital named by S.Botkin, Moscow
  - Federal Almazov North-West Medical Research Centre, Saint Petersburg

REFERENCES:
- [Result] Mian AA, Rafiei A, Haberbosch I, Zeifman A, Titov I, Stroylov V, Metodieva A, Stroganov O, Novikov F, Brill B, Chilov G, Hoelzer D, Ottmann OG, Ruthardt M. PF-114, a potent and selective inhibitor of native and mutated BCR/ABL is active against Philadelphia chromosome-positive (Ph+) leukemias harboring the T315I mutation. Leukemia. 2015 May;29(5):1104-14. doi: 10.1038/leu.2014.326. Epub 2014 Nov 14. PMID 25394714
- [Derived] Turkina A, Vinogradova O, Lomaia E, Shatokhina E, Shukhov O, Chelysheva E, Shikhbabaeva D, Nemchenko I, Petrova A, Bykova A, Siordiya N, Shuvaev V, Mikhailov I, Novikov F, Shulgina V, Hochhaus A, Ottmann O, Cortes J, Gale RP, Chilov G. Phase-1 study of vamotinib (PF-114), a 3rd generation BCR::ABL1 tyrosine kinase-inhibitor, in chronic myeloid leukaemia. Ann Hematol. 2025 May;104(5):2707-2715. doi: 10.1007/s00277-025-06239-8. Epub 2025 Apr 29. PMID 40298994
- See also: doi:10.1038/leu.2014.326 — http://www.nature.com/leu/journal/v29/n5/full/leu2014326a.html